CLINICAL TRIAL: NCT07358273
Title: Conservative Care Versus Decompression Trial for Degenerative Cervical Myelopathy Pilot: A Multicenter Randomized Controlled Feasibility Trial
Brief Title: Conservative Care Versus Decompression Trial for Degenerative Cervical Myelopathy Pilot
Acronym: CADET-DCM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5512
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Cervical Myelopathy
Keywords: myelopathy; spinal cord diseases; surgery; conservative care; spine
MeSH Terms: conditions — Spinal Cord Diseases | interventions — Laminectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative Care (Active Comparator): Standard of care intervention
  Interventions: Other: Conservative Care
- Surgical Decompression (Active Comparator): Standard of care intervention
  Interventions: Procedure: Decompression Surgery

INTERVENTIONS:
Procedure: Decompression Surgery — Surgical decompression of the cervical spine
  Arms: Surgical Decompression
Other: Conservative Care — Conservative care Program for cervical myelopathy
  Arms: Conservative Care

SUMMARY:
This study is a pilot randomized clinical trial designed to test whether it is feasible to conduct a larger study comparing two standard treatments for mild degenerative cervical myelopathy (DCM).

The main questions it aims to answer are:

* Can enough participants be recruited and successfully complete follow-up assessments?
* Will participants adhere to their assigned treatment?

Researchers will compare two groups:

* Surgical group: Participants receive decompressive spine surgery (with or without fusion).
* Conservative care group: Participants follow a structured program that includes education, fall prevention strategies, and tailored exercises.

Participants will:

* Complete baseline and follow-up assessments at 6 weeks, 6 months, and 12 months.
* In the surgical group: undergo surgery within 12 weeks of randomization and receive standard post-operative care.
* In the conservative care group: follow a 6-week progressive exercise program and continue self-management strategies.
* Complete a monthly online symptom monitoring questionnaire

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Show evidence of spinal cord compression between C2 and T1 on MRI or CT myelography conducted within 2 years of enrollment
* Present with mild DCM defined as a score of 15-17 on the modified Japanese Orthopaedic Association (mJOA) score

Exclusion Criteria:

* Clinical suspicion that myelopathic symptoms are exacerbated or caused by another neurologic condition (i.e. amyotrophic lateral sclerosis, multiple sclerosis, syringomyelia, peripheral neuropathy)
* Demonstrate ossification of the posterior longitudinal ligament (OPLL)
* Previous cervical spine surgery
* Report known or suspected tandem symptomatic thoracic or lumbar spinal stenosis
* Present with an acute traumatic spinal cord injury (i.e., central cord syndrome)
* Have a prior history of an acute spinal cord injury
* Have spinal cord compression due to an infectious or oncologic process
* Inflammatory arthritis
* Significant active health-related comorbidity (ASA Class IV or higher)
* English language ability insufficient to complete outcome questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Consent proportion | Enrollment
  Total number of participants randomized/ total number of patients approached
Follow-up completion | 6 month follow-up
  Number of participants with 6-month follow up completed/ number of participants randomized
Adherence to intervention | 6 months after enrollment
  Number of participants who proceed with allocated intervention/ number of participants randomized

SECONDARY OUTCOMES:
Patient-derived Modified Japanese Orthopaedic Association Scale (P-mJOA) | Baseline, 6 months, 12 months
  Patient reported outcome assessing (i) upper extremity sensation, (ii) upper extremity motor function, (iii) lower extremity motor function, and (iv) sphincter function. It is used to grade DCM severity, and scored between 0 and 18. Scores of 18 indicate no dysfunction, 15 to 17 indicate mild DCM, 12 to 14 indicate moderate DCM, 11 and lower indicating severe DCM.
Cervical Myelopathy Severity Index (CMSI) | Baseline, 6 months, 12 months
  The Cervical Myelopathy Severity Index (CSMI) assesses neurological function. It is a patient-completed 14-item measure for patients with DCM to evaluate symptom severity and functional limitations. Items span dexterity, balance/gait, pain, sensory impairment, and sphincter dysfunction. Each item is rated on a 4-point scale, from 0 (no difficulty), to 3 (severe difficulty). Total scores range from 0-42, with a higher score indicating higher DCM severity.
Neck Disability Index (NDI) | Baseline, 6 months, 12 months
  The NDI is a continuous measure ranging from 0 to 100 with higher scores indicating more severe disability.
Arm and Shoulder Pain | Baseline, 6 months, 12 months
  This will be measured using the 11-point Numerical Rating Scale (NRS), where 0 is 'no pain' and 10 is 'worst possible pain'.
Upper Extremity Neurologic Function | Baseline, 6 months, 12 months
  This will be measured using the grip-and-release test (G&R test). Participants are asked to grip and release with the fingers as rapidly as possible with the forearm kept in pronation and the wrist in mild extension. The number of complete cycles of movement within 10 seconds are counted.
Lower Extremity Neurologic Function | Baseline, 6 months, 12 months
  This will be measured using the 30-m walking test (30MWT). Participants are asked to walk a straight 30-meter distance as quickly as possible with any normally used walking aids; number of steps and time is recorded.
Falls | Baseline, 6 months, 12 months
  Falls will be assessed using questions one and two of the modified American Geriatric/British Geriatric tool: "How many times have you fallen since the last visit?" and "Since the last visit, did you seek medical care for a fall injury?"
Dysphagia | Baseline, 6 months, 12 months
  Dysphagia will be assessed using the Bazaz Scoring System. This classifies patient reported swallowing difficulty into 4 categories: none, mild, moderate, severe.
Need for additional cervical spine surgery | Up to 12 months after the intervention.
  This will be assessed and collected from patient self-report and medical records.
Adverse Events | Through study completion, up to 12 months after intervention.
  Occurrence of related adverse events will be monitored at every scheduled and unscheduled clinic visit.